CLINICAL TRIAL: NCT02702843
Title: Efficacy Of Near Infrared Incisionless Fluorescent Cholangiography (NIFC) During Laparoscopic Cholecystectomy
Brief Title: Fluorescent Cholangiography vs White Light for Bile Ducts Identification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Cedars-Sinai Medical Center (Other); Tokyo Medical University (Other); Asklepios Kliniken Hamburg GmbH (Other); Università degli Studi dell'Insubria (Other); University of Rostock (Other); Hospital de Clinicas José de San Martín (Other)
Responsible Party: Principal Investigator, Emanuele LoMenzo, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FLA 15-108
Record Dates: First submitted 2016-02-17; First posted 2016-03-09 (Estimated); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Cholecystitis; Cholelithiasis
MeSH Terms: conditions — Cholecystitis; Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xenon Light (Active Comparator): Laparoscopic cholecystectomy with Xenon Light
  Interventions: Procedure: Laparoscopic cholecystectomy with Xenon light
- Near infrared light (Experimental): Laparoscopic cholecystectomy with Near infrared light
  Interventions: Procedure: Laparoscopic cholecystectomy with Xenon light; Procedure: Laparoscopic cholecystectomy (fluorescent cholangiography)

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy with Xenon light — Standard laparoscopic cholecystectomy with white light
Procedure: Laparoscopic cholecystectomy (fluorescent cholangiography) — Laparoscopic cholecystectomy in infrared light after injection of indocyanine green pre-operatively.
  Arms: Near infrared light

SUMMARY:
The Study is designed to compare the effectiveness of Near Infrared Fluorescence Cholangiography (NIFC) to standard white light imaging (WLI) in visualizing and identifying the main biliary and hepatic structures (Cystic Duct, Right Hepatic Duct, Common Hepatic Duct, Common Bile Duct, Cystic-CBD junction, Cystic-Gallbladder junction and any Accessory Ducts) during laparoscopic cholecystectomy. The aim is to demonstrate that NIFC performs better than standard white light (WLI) alone in visualizing and identifying extra-hepatobiliary structures (Cystic Duct, Right Hepatic Duct, Common Hepatic Duct, Common Bile Duct, Cystic-CBD junction, Cystic-Gallbladder junction, and any Accessory Ducts) before and after dissection during Laparoscopic Cholecystectomy (LC).

DETAILED DESCRIPTION:
Recently, a novel technique to visualize structures using fluorescent light and intravenous dye has been developed.

Near Infrared Incisionless Fluorescent Cholangiography (NIFC) is a medical imaging technique that uses fluorescence to detect properly labeled structures during surgery.

NIFC is performed using imaging devices with the purpose of providing real-time simultaneous information from color reflectance images (white light) and fluorescence emission (near infrared light). One or more light sources are used to excite and illuminate the sample. Light is collected using optical filters that match the emission spectrum of the fluorophore. Imaging lenses and digital cameras are used to produce the final image.

During laparoscopic cholecystectomies, the visualization of the extra-hepatic bile ducts with fluorescence is called Near Infrared Incisionless Fluorescent Cholangiography (NIFC). Fluorescence equipment and a dye are necessary in order to perform a NIFC, but the technique requires no radiation or incision. A fluorescence dye is administrated intravenously at least 45 minutes before the surgery, which is excreted by the liver and the bile duct The Study is designed to compare the effectiveness of Near Infrared Fluorescence Cholangiography (NIFC) to standard white light imaging (WLI) in visualizing and identifying the main biliary and hepatic structures (Cystic Duct, Right Hepatic Duct, Common Hepatic Duct, Common Bile Duct, Cystic-CBD junction, Cystic-Gallbladder junction and any Accessory Ducts) during laparoscopic cholecystectomy.

Eligible patients will be identified through clinical and test evaluation. Eligibility will be verified by the patient's primary surgeon. The surgeon will determine the indication and date of the surgery. Once a patient is confirmed as eligible, the surgeon will introduce the study in detail. If after being introduced to the study and having had the opportunity to ask questions, the patient is willing to participate, he/she will be asked to review and sign the informed consent document .

Upon entry in the clinical trial patients will be randomly allocated to the intervention arm. Data will be collected at enrolment time, during surgery, at the end of surgery and one week after surgery.

Upon entry in the clinical trial, the master study database (REDCap, will randomly allocated patients to one of the study arms (1:1) within site (1:1) using a computer generated random sequence. This will provide an allocation sequence for each site. Once a patient is enrolled and a database file in REDCap is initiated for that patient, he/she will be assigned electronically to one of the study arms.

Patient will be blind to the intervention but surgeon blinding will not be feasible due to the nature of the intervention. The study will involve a considerable number of surgeons in each site, which should compensate any potential bias of some of them in favor or against either approach.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders
2. Minimum age: 18 years old
3. Spoken and written command of the language spoken in the country's center
4. Ability to understand and follow the study procedures and sign the informed consent

Exclusion Criteria:

1. Known allergies to iodides
2. Known history of coagulopathy
3. Known moderate or severe liver disease Women who are pregnant or breastfeeding, or for whom possibility of pregnancy was not ruled out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Rosenthal, MD, Principal Investigator — Cleveland Clinic Florida
Locations (7):
- United States (2):
  - Cedar Sinai, Los Angeles, California
  - Cleveland Clinic, Cleveland, Ohio
- Hospital de clinicas jose de San Martin, Buenos Aires, Argentina
- Germany (2):
  - Askelopios Westklinikum Hamburg, Hamburg
  - Klinikum Sudstadt Rostock, Rostock
- University of Insubria, Varese, Italy
- University of Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Redcap will be used Data to be shared - pre-operative data including age, sex, laboratory values and imaging, intra-operative data including visualization of the extra-hepatic biliary structure with white light and with infrared light by the operating surgeon and the observer, any bile leak; post-operative data documenting any complications such as reaction to ICG or bile duct injury.
  Data will be available as each center finishes up the follow of each individual patient (usually 2 weeks post operatively). Each center will update the data on Redcap on a monthly basis.
  Data will be initially obtained on a pre-decided forms (approved by the IRB committee) and transferred to Redcap for electronic record keeping and analysis.

REFERENCES:
- [Derived] Dip F, LoMenzo E, Sarotto L, Phillips E, Todeschini H, Nahmod M, Alle L, Schneider S, Kaja L, Boni L, Ferraina P, Carus T, Kokudo N, Ishizawa T, Walsh M, Simpfendorfer C, Mayank R, White K, Rosenthal RJ. Randomized Trial of Near-infrared Incisionless Fluorescent Cholangiography. Ann Surg. 2019 Dec;270(6):992-999. doi: 10.1097/SLA.0000000000003178. PMID 30614881

RESULTS

PARTICIPANT FLOW:
Groups:
- Near Infrared Light: Laparoscopic cholecystectomy with Near infrared light
  Laparoscopic cholecystectomy with Xenon light: Standard laparoscopic cholecystectomy with white light
  Laparoscopic cholecystectomy (fluorescent cholangiography): Laparoscopic cholecystectomy in infrared light after a single injection of 5 cc of indocyanine green at least 30 minutes pre-operatively.
Period: Overall Study
Arm/Group | Xenon Light | Near Infrared Light
Started | 333 | 344
Completed | 318 | 321
Not Completed | 15 | 23
Not completed — Insufficient data to analyze | 15 | 23

BASELINE CHARACTERISTICS:
Population: All participants who completed the study procedures and had available documentation were included in the baseline analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Xenon Light | Near Infrared Light | Total
Number analyzed (Participants) | 318 | 321 | 639
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 261 | 264 | 525
  >=65 years | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (15.5) | 48.3 (15.0) | 48.4 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 218 | 399
  Male | 137 | 103 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 318 | 321 | 639
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 318 | 321 | 639
Region of Enrollment [Number; unit: participants]
  Argentina | 96 | 104 | 200
  United States | 83 | 74 | 157
  Japan | 0 | 1 | 1
  Italy | 33 | 31 | 64
  Germany | 106 | 111 | 217

OUTCOME MEASURES:

1. Primary Outcome: Detection Rate of Common Bile Duct Before and After Dissection Using Near Infra-red Light
Description: Detection rate of the common bile duct during laparoscopic cholecystectomy, defined as the proportion of patients in whom the common bile duct was visualized immediately before dissection (baseline) and immediately after dissection using near infrared light. The detection rate was calculated separately for each arm and reported as the percentage of patients with successful identification.
Time Frame: Immediately before dissection (baseline) and immediately after dissection during the same surgical procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Xenon Light | Near Infrared Light
Number analyzed (Participants) | 318 | 321
Participants
  Before Dissection | 64 | 157
  After Dissection | 159 | 243

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Xenon Light | Near Infrared Light
All-Cause Mortality (participants affected / at risk) | 1/318 | 0/321
Serious Adverse Events (participants affected / at risk) | 2/318 | 0/321
Other Adverse Events (participants affected / at risk) | 4/318 | 1/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xenon Light (N=318) | Near Infrared Light (N=321)
Bile Duct Injury (Hepatobiliary disorders) | 2 (2) | 0 (0) — Intraoperative Common Bile Duct Injury
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xenon Light (N=318) | Near Infrared Light (N=321)
Conversion to Open (Surgical and medical procedures) | 4 (4) | 1 (1) — Conversion from laparoscopy to laparotomy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT02702843/Prot_SAP_ICF_000.pdf